CLINICAL TRIAL: NCT05715086
Title: Upfront vs Postponed Ureteroscopy (UPURS) Trial for Patient-centered Management of Symptomatic Obstructing Stones
Brief Title: UPURS Trial for Patient-centered Management of Symptomatic Obstructing Stones
Acronym: UPURS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Colorado, Denver (Other); State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-37665
Record Dates: First submitted 2022-12-16; First posted 2023-02-06 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Ureteral Stone
Keywords: Symptomatic ureteral stones
MeSH Terms: conditions — Ureterolithiasis | interventions — Ureteroscopy

STUDY DESIGN:
Intervention Model Description: A prospective, non-blinded, randomized controlled trial with two study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Upfront ureteroscopy) (Active Comparator)
  Interventions: Procedure: Ureteroscopy
- Group B (Observation/delayed ureteroscopy) (No Intervention)

INTERVENTIONS:
Procedure: Ureteroscopy — Upfront ureteroscopy
  Arms: Group A (Upfront ureteroscopy)

SUMMARY:
A prospective, non-blinded, randomized controlled trial studying the management of symptomatic ureteral stones. This study will compare upfront ureteroscopy vs observation and delayed intervention for patients presenting to the emergency department with a symptomatic ureteral stone.

DETAILED DESCRIPTION:
Management of symptomatic ureteral stones is variable across the United States due to a lack of clear, patient-centered guidelines. For patients who do not meet criteria for emergent stenting, the decision to recommend upfront definitive treatment (ureteroscopy, ESWL) or medical expulsion therapy is influenced by factors such as practice setting, insurance status, and day of the week. This has resulted in health disparities and delays in care that disproportionately affect vulnerable patient populations.

For patients presenting to the emergency department with a symptomatic ureteral stone investigators will randomize into Group A: Upfront Ureteroscopy or Group B: Delayed intervention and observation. Both arms are considered standard of care for patients presenting with the above diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to the Emergency Department (ED)
* Adult (> 18 yo)
* ≥5mm ureteral stone diagnosed on CT scan
* Presence of symptoms (pain, nausea, vomiting, hematuria)

Exclusion Criteria:

* Strict indication for stent
* Stone burden not amenable to Ureteroscopy (URS)
* Dirty urine analysis (UA) or positive urine culture (UCx)
* Transplant kidney
* Presence of conduit
* Comorbidities not optimized for surgery
* Strong preference for surgery or observation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 3 months
  Measure on a scale of 1-10, with zero indicating no pain and 10 indicating the worst pain.
Anxiety Score | 3 months
  Measure on a scale of 1-10, the score ranges from 0-10, with zero indicating no anxiety and 10 indicating the worst anxiety.

SECONDARY OUTCOMES:
Hospital visit length | 3 months
  Measured in number of days

OTHER OUTCOMES:
Days of work lost | 3 months
  Measured in number of days
Hospital visits | 3 months
  Measure in number of times

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Chi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No